CLINICAL TRIAL: NCT04475900
Title: Computer-aided Diagnosis of Ocular Diseases Based on Corneal Biomechanics - Selection and Evaluation of Eligible Patients With Certain Ocular Diseases Associated With Biomechanical Alterations
Brief Title: Computer-aided Diagnosis of Ocular Diseases Based on Corneal Biomechanics
Acronym: EyeTwin
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: Fraunhofer Institute for Ceramic Technologies and Systems IKTS (Unknown)
Responsible Party: Sponsor
Other Study IDs: BO-EK-195052020
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Corneal Ectasia; Corneal Disease; Corneal Astigmatism; Keratoconus; Glaucoma; Open Angle Glaucoma; Normal Tension Glaucoma
Keywords: Cornea; Ectasia; Keratoconus; Finite Element Modelling; computer-aided data analysis; Glaucoma; Corneal biomechanics
MeSH Terms: conditions — Corneal Diseases; Astigmatism; Keratoconus; Glaucoma; Glaucoma, Open-Angle; Low Tension Glaucoma; Dilatation, Pathologic | interventions — Vision, Ocular; Corneal Topography; Tomography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Healthy: Healthy eyes without any signs of ocular diseases
  Interventions: Diagnostic Test: Corneal biomechanics (Corvis ST, Oculus, Wetzlar, Germany); Diagnostic Test: Corneal topography and tomography (Pentacam, Oculus, Wetzlar, Germany); Diagnostic Test: Optic nerve head measurement
- Ectasia: ectasia suspects early, moderate and advanced keratoconus
  Interventions: Diagnostic Test: Corneal biomechanics (Corvis ST, Oculus, Wetzlar, Germany); Diagnostic Test: Corneal topography and tomography (Pentacam, Oculus, Wetzlar, Germany)
- Glaucoma: Normal Tension glaucoma Primary Open-Angle Glaucoma
  Interventions: Diagnostic Test: Corneal biomechanics (Corvis ST, Oculus, Wetzlar, Germany); Diagnostic Test: Corneal topography and tomography (Pentacam, Oculus, Wetzlar, Germany); Diagnostic Test: Optic nerve head measurement

INTERVENTIONS:
Diagnostic Test: Corneal biomechanics (Corvis ST, Oculus, Wetzlar, Germany) — To measure corneal biomechanics with Scheimpflug based tonometry
Diagnostic Test: Corneal topography and tomography (Pentacam, Oculus, Wetzlar, Germany) — To measure corneal topography and tomography with Scheimpflug tomograph
Diagnostic Test: Optic nerve head measurement — To measure optic nerve excavation
  Groups: Glaucoma; Healthy

SUMMARY:
The purpose of this study is the investigation of biomechanical properties of the cornea using computer-aided data analysis. Currently, it is known that keratoconus and glaucoma are ocular disease that are associated with biomechanical alterations of the cornea. Corneal ectasia, especially keratoconus, is a corneal disease that leads to an irreversible loss of visual acuity while the cornea becomes steeper, thinner and irregular. For these patients, surgical intervention (e.g. corneal cross-linking) is performed, in case of disease progression. In glaucoma, the information about corneal alterations serves in two ways, first, correct measurement of intra ocular pressure (IOP); second, early diagnosis of suspects before visual field defects are detectable.

Especially, the Corvis ST is an air-puff tonometer that measures intraocular pressure, corneal thickness (CCT) as well as dynamic corneal response (DCR) parameters. Most of the DCR parameters are affected by IOP and CCT: Therefore, algorithm are needed to determine parameters without impact of IOP and CCT that are describe the biomechanical properties of the cornea.

DETAILED DESCRIPTION:
In this study, an eye twin based on finite element modeling is used to measure advanced properties of corneal biomechanics. Raw data of Corvis ST measurement are exported from the device and imported into the model. The outcome of these calculations are merged together and are compared to further clinical findings (e. g. corneal topography and tomography, axial eye length).

Further information were obtained:

Age, sex, refraction, family history, known duration of disease, previous ocular surgery, systemic diseases, systemic and topical medication; biomicroscopy, anterior optical coherence tomography (OCT), Scheimpflug-based tomography (Pentacam), Biomechanical assessment (Ocular Response Analyzer and Corneal Visualization with the Scheimpflug Technology), optical biometry, confocal microscopy, endothelium cell count.

ELIGIBILITY:
Inclusion Criteria:

* corneal ectasia (keratoconus) or ectasia suspect
* glaucoma (Primary open angle glaucoma and normal Tension glaucoma) or glaucoma suspect

Exclusion Criteria:

* age under 18 years
* pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with corneal ectasia or glaucoma. Healthy eyes that matching to ocular disease groups concerning age.
Sampling Method: Probability Sample
Enrollment: 372 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
New biomechanical parameters of the cornea | 2 years
  To detemine biomechanical alterations in different ocular diseases and correlate them with other clinical findings

SECONDARY OUTCOMES:
Dependence of new biomechanical Parameters of the cornea from influencing factors | 1 year
  e. g. corneal thickness, intraocular pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology; Medical Faculty Carl Gustav Carus; Technical University Dresden, Dresden, Saxony, Germany